CLINICAL TRIAL: NCT03872531
Title: Lifetime Impact Study for Achondroplasia (LISA)
Brief Title: Lifetime Impact Study for Achondroplasia
Acronym: LISA
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 111-502
Record Dates: First submitted 2019-01-16; First posted 2019-03-13 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Cohort 1: Includes age group 3-5 with a cap at 20 subjects. This is a retrospective, observational study
- Cohort 2: Includes age group 6-10 with a cap at 30 subjects. This is a retrospective, observational study
- Cohort 3: Includes age group 11-15 with a cap of 30 subjects. This is a retrospective, observational study
- Cohort 4: Includes age group 16-20 with a cap of 20 subjects. This is a retrospective, observational study
- Cohort 5: Includes age group 21-30 with a cap at 20 subjects. This is a retrospective, observational study
- Cohort 6: Includes age group 31-40 with a cap at 20 subjects. This is a retrospective, observational study
- Cohort 7: Includes age group 41 and over with a cap at 35 subjects. This is a retrospective, observational study

SUMMARY:
Observational study looking at the burden of illness in achondroplasia subjects aged 3 and above. The study will include a 3 year review of historical clinical data as well as a single point collection of questionnaire data to look at the impact on the following in individuals with achondroplasia versus a normative population:

* Quality of life
* Clinical burden
* Healthcare resource use
* Socio-economic burden
* Psychosocial burden

Up to 175 subjects will be enrolled in sites in Argentina, Colombia and Brazil.

DETAILED DESCRIPTION:
This is a multinational, epidemiological, observational, retrospective, cross-sectional study of individuals with achondroplasia (subjects). This study will be conducted at up to approximately 4 sites in Latin American Countries - Brazil, Argentina and Colombia.

Subjects will be identified for participation in the study via three routes:

1. During routine hospital visits
2. From clinic lists of those previously treated but no longer followed at the study site.
3. Through collaboration of the Investigator with Achondroplasia patient organizations, other Achondroplasia-related organizations, other healthcare professionals in their country and Achondroplasia-related social media sites. A recruitment flyer will be provided to these organizations, healthcare professionals and distributed to potential subjects.

Data will be collected over a minimum of the three years prior to the date of enrolment. Clinical and healthcare resource use data will be collected from medical records. For each subject enrolled, data from medical records will be collected and entered onto an electronic case report form (eCRF) at each site. Data collection from medical records will be supplemented by records provided by the subject and, if necessary, confirmed by the family Doctor.

Data about QoL, mobility, psychosocial burden, socio-economic burden and healthcare resource use will be collected via a booklet of validated and structured questionnaires.

Characteristics of subjects with achondroplasia (QoL scores, healthcare resource use, educational level, family status, employment status) will be compared with those of the general population, where available.

As this is an observational study, participation will not affect the subject/Investigator relationship, nor influence Investigator's treatment, therapeutic or other management of the subject.

Subject participation onto the study will be voluntary, without financial support to the subject.

ELIGIBILITY:
Inclusion Criteria:

1. Individual with a documented diagnosis of achondroplasia based on:

   1. Genetic confirmation of achondroplasia and/or
   2. Clinical diagnosis of achondroplasia (clinical examination and/or radiological assessment)
2. ≥ three years of age at the time of enrollment
3. Has the cognitive and linguistic capacities necessary to complete questionnaires in the language of his/her country (and/or parents/legally acceptable representatives, as applicable)
4. Agrees to participate in the study and has read, understood, completed and signed:

   1. Informed Consent Form (ICF) - for adult subjects
   2. Informed Assent Form (IAF) - for minor subjects, accompanied by a parental ICF completed by their parents/legally acceptable representatives. The age at which the minor subjects sign the IAF will be subject to local requirements.
5. Has medical records available for the three years prior to the date of enrollment.

Exclusion Criteria:

1. Currently participating, or participated in the last six months, in

   1. a clinical trial of a medicinal product or medical device or
   2. other non-clinical or low interventional studies
2. Currently participating or has participated in any BioMarin study at any time.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of Achondroplasia aged 3 years or older in Argentina, Brazil and Colombia
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Healthcare resource use | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  Healthcare resource use will be collected from medical records and through patient questionnaires. Data collection from medical records will be supplemented by records provided by the subject and, if necessary, confirmed by the family doctor. Healthcare resource use will be collected via validated and structured questionnaires

SECONDARY OUTCOMES:
Socio-economic burden | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  Data about socio-economic burden will be collected via validated and structured questionnaires specifically the Work and Productivity and Activity Impairment (WPAI-SHP)
Pediatric Functional Independence Measure (WeeFIM) | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  The WeeFIM measures the need for assistance and the severity of disability in children between six months and seven years of age. The instrument consists of 18 items covering three domains: self-care, mobility, and cognition. The mean total score within each domain and the overall total score will be summarized. The study will be assessing subjects aged from 3 to 17 years
Adolescent Pediatric Pain Tool (APPT) | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  The APPT is an instrument for self-reporting of pain by children and adolescents aged 8-17 years. Five subscale scores will be summarized on the analysis population
Pediatric Quality of Life Inventory (PedsQL) | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  The PedsQL is comprised of four dimensions: Physical, Emotional, Social, and School Functioning. The overall score for each dimension is defined as the mean score for each item involved in the dimension. The overall score for each dimension and the mean total score across dimensions will be summarized for each report.
Quality of Life Short Stature Youth (QoLiSSY) Questionnaire | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  The QoLISSY Questionnaire for children and adolescents consists of the core QOL dimensions: Physical, Social and Emotional, and three predictors of quality of life: Coping, Beliefs and Treatment. The QoLISSY total score is calculated by the sum of the means in the physical, social and emotional sub-scales divided by 3.
Nottingham Health Profile(NHP) Questionnaire | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  The NHP is a generic quality of life survey used to measure subjective physical, emotional, and social aspects of health. The NHP total score is calculated by averaging the six domain scores.
Brief Pain Inventory-Short Form (BPI-SF) Questionnaire | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  The BPI-SF is used to assess clinical pain. A mean severity score and mean interference score will be calculated and summarized for the analysis population
EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) Questionnaire | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  EQ-5D-5L questionnaire has 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 5 problem levels corresponding to patient response choices. A quality of life score is obtained according to the answers to the questionnaires.
Child Behaviour Checklist (CBCL) | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  The CBCL questionnaire is completed by the parent to assess the child behavioral and emotional problems. The questions are grouped into eight categories which focus on different aspects of behavior: aggressive behavior, anxious/depressed, attention problems, rule-breaking behavior, somatic complaints, social problems, thought problems and withdrawn/depressed.
Understanding the Impact of Achondroplasia on Quality of Life Questionnaire | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at end of study with the final Clinical Study Report, May 2020
  Impact on anxiety, depression, sleep disturbance and impact on relationships with others (spouse/partner family members, friends), social life and activities, perception of health, self-esteem, plans/ambitions for the future.

OTHER OUTCOMES:
Measurement of Height | Retrospective data will be collected for 3 years prior to date of enrolment
  Height measurements will be collected from retrospective data where available for standing and sitting height measurements. The height data will be measured in centimetres.
Measurement of Weight | Retrospective data will be collected for 3 years prior to date of enrolment
  Weight will be collected from retrospective data collected and will be entered in kilograms.
Body Mass Index (BMI) | Retrospective data will be collected for 3 years prior to date of enrolment
  Body Mass Index is calculated using height and weight. Body Mass Index (BMI) will be measured in kg/m2
Head Circumference | Retrospective data will be collected for 3 years prior to date of enrolment
  Head Circumference will be collected from retrospective data collected and will be entered in centimetres.
Upper and Lower Arm Length | Retrospective data will be collected for 3 years prior to date of enrolment
  Upper and Lower Arm Length will be collected from retrospective data collected and will be entered in centimetres.
Iliac Height (hip to floor) | Retrospective data will be collected for 3 years prior to date of enrolment
  Iliac Height (hip to floor) will be collected from retrospective data collected and will be entered in centimetres.
Subischial Length | Retrospective data will be collected for 3 years prior to date of enrolment
  Subischial Length will be collected from retrospective data collected and will be entered in centimetres.
Thigh Length | Retrospective data will be collected for 3 years prior to date of enrolment
  Thigh Length will be collected from retrospective data collected and will be entered in centimetres.
Knee Height | Retrospective data will be collected for 3 years prior to date of enrolment
  Knee Height will be collected from retrospective data collected and will be entered in centimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — BioMarin Pharmaceutical
Locations (4):
- Hospital de Pediatría "Prof. Dr. Juan P. Garrahan", Buenos Aires, Argentina
- Brazil (2):
  - Instituto Nacional Fernandes Figueira (IFF), Fundacao Osvaldo Cruz, Rio de Janeiro
  - Centro de Pesquisa Clínica do Instituto da Criança HC - FMUSP, São Paulo
- Fundacion Cardioinfantil-instituto de cardiologia, Bogotá, Colombia